CLINICAL TRIAL: NCT00176345
Title: Impact of Exercise Training on Bradykinin-Mediated Endothelial Function in Patients With Coronary Artery Disease
Brief Title: Impact of Exercise Training on Endothelial Function in CAD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leipzig (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 639/97; 157/02
Record Dates: First submitted 2005-09-11; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-09

CONDITIONS: Coronary Artery Disease
Keywords: exercise training; endothelial function
MeSH Terms: conditions — Coronary Artery Disease | interventions — Exercise

INTERVENTIONS:
Behavioral: Exercise Training

SUMMARY:
Bradykinin has been identified to contribute to the release of nitric oxide (NO), prostacyclin, and EDHF through activation of specific bradykinin 2 (B2) receptors, which is finally promoting a vasodilatory respone. Regular physical exercise training results in an improvement of endothelial function in patients with CAD. These positive effects were partially attributed to an increased expression of endothelial NO synthase (eNOS) and cyclooxygenase (COX) as a result of the training intervention.

Aim of this trial is therefore to determine, whether the training-induced correction of endothelial dysfunction is also bradykinin-dependent.

DETAILED DESCRIPTION:
A total of 20 patients with stable coronary artery disease are prospectively randomized to 4 weeks of exercise training or sedentary lifestyle.

Endothelial function of the radial artery is determined by a high-resolution A-mode ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* stable CAD
* male gender

Exclusion Criteria:

* insulin-dependent diabetes mellitus
* significant valvular heart disease
* smoking
* exercise-induced myocardial ischemia
* conditions prohibiting exercise training

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2001-01

PRIMARY OUTCOMES:
Endothelial function

CONTACTS AND LOCATIONS:
Overall Officials: Rainer P Hambrecht, MD, Principal Investigator — University of Leipzig, Heart Center, Department of Internal Medicine / Cardiology
Locations (1):
- University of Leipzig, Heart Center, Department of Internal Medicine / Cardiology, Leipzig, Saxony, Germany